CLINICAL TRIAL: NCT02511210
Title: Comparison of the Effects of Regional Anesthesia / Peripheral Nerve Block and General Anesthesia on Preoperative Anxiety
Brief Title: Regional Anesthesia / Peripheral Nerve Block and General Anesthesia on Preoperative Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Collaborators: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, M.D, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: erzincan university
Record Dates: First submitted 2015-07-24; First posted 2015-07-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-09

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Anesthesia, Conduction; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- regional anesthesia (Active Comparator): spinal anesthesia or peripheral nerve block
  Interventions: Behavioral: regional anesthesia
- general anesthesia (Active Comparator): intubated patients
  Interventions: Behavioral: general anesthesia

INTERVENTIONS:
Behavioral: regional anesthesia — preoperative anxiety
  Arms: regional anesthesia
Behavioral: general anesthesia — preoperative anxiety
  Arms: general anesthesia

SUMMARY:
The researchers aimed to investigate that preoperative anxiety scores of patients who are informed about the anesthesia before surgery with using State-Trait Anxiety Inventory and Amsterdam preoperative anxiety and information scale tests together.

DETAILED DESCRIPTION:
Patients will be informed about the anesthesia procedure in service ad then It will be held anxiety questionnaires one day before surgery and operation rooms.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80,
* both women and men,
* Patients will be operated

Exclusion Criteria:

* psychiatric and neurologic diseases,
* hearing and speech disorders,
* Psychiatric drug and chronic alcohol use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory scores in patients undergoing regional anesthesia | two months

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory scores in operating rooms | two months
Amsterdam Preoperative Anxiety and Information Scale scores in operating rooms | two months
Amsterdam Preoperative Anxiety and Information Scale scores in patients undergoing regional anesthesia | two months

CONTACTS AND LOCATIONS:
Overall Officials: ILKE KUPELI, M.D, Principal Investigator — Erzincan University
Locations (1):
- Mengucek Gazi Training and Research Hospital, Erzincan, Merkez, Turkey (Türkiye)

REFERENCES:
- [Background] Perks A, Chakravarti S, Manninen P. Preoperative anxiety in neurosurgical patients. J Neurosurg Anesthesiol. 2009 Apr;21(2):127-30. doi: 10.1097/ANA.0b013e31819a6ca3. PMID 19295391
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Caumo W, Schmidt AP, Schneider CN, Bergmann J, Iwamoto CW, Adamatti LC, Bandeira D, Ferreira MB. Risk factors for postoperative anxiety in adults. Anaesthesia. 2001 Aug;56(8):720-8. doi: 10.1046/j.1365-2044.2001.01842.x. PMID 11493233
- [Background] Markland D, Hardy L. Anxiety, relaxation and anaesthesia for day-case surgery. Br J Clin Psychol. 1993 Nov;32(4):493-504. doi: 10.1111/j.2044-8260.1993.tb01085.x. PMID 8298547
- [Background] Badner NH, Nielson WR, Munk S, Kwiatkowska C, Gelb AW. Preoperative anxiety: detection and contributing factors. Can J Anaesth. 1990 May;37(4 Pt 1):444-7. doi: 10.1007/BF03005624. PMID 2340614
- [Background] Kain ZN, Kosarussavadi B, Hernandez-Conte A, Hofstadter MB, Mayes LC. Desire for perioperative information in adult patients: a cross-sectional study. J Clin Anesth. 1997 Sep;9(6):467-72. doi: 10.1016/s0952-8180(97)00102-5. PMID 9278833
- [Background] Kain ZN, Wang SM, Caramico LA, Hofstadter M, Mayes LC. Parental desire for perioperative information and informed consent: a two-phase study. Anesth Analg. 1997 Feb;84(2):299-306. doi: 10.1097/00000539-199702000-00011. PMID 9024018
- [Background] Tenenbaum G, Furst D, Weingarten G. A statistical reevaluation of the STAI anxiety questionnaire. J Clin Psychol. 1985 Mar;41(2):239-44. doi: 10.1002/1097-4679(198503)41:23.0.co;2-5. PMID 3980747
- [Result] Spielberger CD, Auerbach SM, Wadsworth AP, Dunn TM, Taulbee ES. Emotional reactions to surgery. J Consult Clin Psychol. 1973 Feb;40(1):33-8. doi: 10.1037/h0033982. No abstract available. PMID 4688678
- [Result] Norris W, Baird WL. Pre-operative anxiety: a study of the incidence and aetiology. Br J Anaesth. 1967 Jun;39(6):503-9. doi: 10.1093/bja/39.6.503. No abstract available. PMID 6027959
- [Result] Hicks JA, Jenkins JG. The measurement of preoperative anxiety. J R Soc Med. 1988 Sep;81(9):517-9. doi: 10.1177/014107688808100907. PMID 3184108
- [Result] Johnston M. Anxiety in surgical patients. Psychol Med. 1980 Feb;10(1):145-52. doi: 10.1017/s0033291700039684. PMID 7384316
- [Result] Maheshwari D, Ismail S. Preoperative anxiety in patients selecting either general or regional anesthesia for elective cesarean section. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):196-200. doi: 10.4103/0970-9185.155148. PMID 25948900
- [Result] Deniz Erdem, Cengiz Ugiş, M. Demet Albayrak, Belgin Akan, Esra Aksoy, Nermin Göğüş. Perianal Bölge Ameliyatı Yapılacak Hastalarda Uygulanan Anestezi Yöntemlerinin Preoperatif ve Postoperatif Anksiyete ve Ağrı Düzeylerine Etkisi. Bakırköy Tıp Dergisi 2011;7:11-16